CLINICAL TRIAL: NCT07394738
Title: Evaluating the Effectiveness of Various Biomaterials for Alveolar Socket Preservation
Brief Title: Using Different Biomaterials to Preserve Bone After Tooth Extraction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Okan Ozen, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSA-2024-180
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-04

CONDITIONS: Alveolar Ridge Preservation; Bone Regeneration; Tooth Extraction; Dental Implants
Keywords: Alveolar Socket Preservation; Autogenous Dentin Graft; Socket Healing
MeSH Terms: interventions — Transplantation, Homologous; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Four-arm randomized parallel study comparing allograft, autogenous dentin graft, dentin graft + hyaluronic acid, and natural healing in post-extraction sockets.
Masking Description: Histological evaluator will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Allograft (Experimental): Participants receive an allograft material placed into the extraction socket. Healing and gingival parameters are assessed at predefined time points.
  Interventions: Other: Allograft
- Dentin Graft (Experimental): Participants receive autogenous dentin graft material placed into the extraction socket. Healing and gingival parameters are assessed at predefined time points.
  Interventions: Other: Autogenous Dentin Graft
- Dentin + Hyaluronic Acid (Experimental): Participants receive a combination of autogenous dentin graft and hyaluronic acid placed into the extraction socket. Healing and gingival parameters are assessed at predefined time points.
  Interventions: Other: Autogenous Dentin Graft; Other: Hyaluronic Acid Gel
- Natural Healing (No Intervention): Extraction sockets are left to heal without the application of graft or biomaterial. Healing and gingival outcomes are evaluated at predefined time points.

INTERVENTIONS:
Other: Allograft — Following tooth extraction, the socket is filled with particulate freeze-dried allograft. The material is placed in a single session immediately after extraction to support socket preservation. Healing is monitored clinically at scheduled follow-up visits.
  Other Names: Freeze-dried allograft material
  Arms: Allograft
Other: Autogenous Dentin Graft — After tooth extraction, autogenous dentin is processed into particulate graft form and placed into the socket in the same session. The graft is used for socket preservation, and healing is assessed clinically during planned follow-up visits.
  Other Names: Dentin particulate graft
  Arms: Dentin + Hyaluronic Acid; Dentin Graft
Other: Hyaluronic Acid Gel — A hyaluronic acid gel is applied as an adjunct biomaterial in combination with dentin graft material during socket preservation. Tissue response is evaluated at scheduled follow-up visits.
  Other Names: Hyaluronic acid (HA); HA gel
  Arms: Dentin + Hyaluronic Acid

SUMMARY:
This clinical study aims to evaluate the effectiveness of different biomaterials in alveolar socket preservation following tooth extraction. Participants will be allocated into three groups: (1) dentin graft, (2) dentin graft combined with hyaluronic acid, and (3) natural healing without any grafting material (control group). At 4 months post-extraction, dental implants will be placed, and bone biopsies will be obtained during the procedure. These biopsy samples will be subjected to histological analysis to assess new bone formation and graft integration. The study will contribute to the understanding of biomaterial performance in socket preservation prior to implant placement.

DETAILED DESCRIPTION:
This randomized clinical trial is designed to evaluate the clinical and histological outcomes of different biomaterials used for alveolar socket preservation following tooth extraction. A total of 36 systemically healthy adult patients requiring tooth extraction in the non-molar region will be enrolled and randomly assigned to one of the following three groups (12 patients per group):

Group 1: Extraction socket filled with autogenous dentin graft.

Group 2: Extraction socket filled with autogenous dentin graft combined with hyaluronic acid.

Group 3 (Control): Extraction socket left to heal naturally without any graft material.

All patients will be re-evaluated at 4 months post-extraction, at which time dental implant placement will be performed. During the implant surgery, bone core biopsies will be taken from the grafted sites using a trephine bur for histological analysis. These specimens will be evaluated to assess new bone formation, residual graft material, inflammatory response, and overall bone quality.

Clinical parameters such as soft tissue healing, postoperative complications, and patient-reported outcomes will also be recorded throughout the healing period.

This study aims to compare the regenerative potential of dentin graft and dentin graft combined with hyaluronic acid, and to determine whether these materials can enhance socket healing and improve bone quality prior to implant placement.

ELIGIBILITY:
Inclusion Criteria Adults aged 18 years or older

Indicated for tooth extraction in the anterior or premolar region of the maxilla or mandible

Planned socket preservation and subsequent dental implant placement at the extraction site

Adequate bone volume permitting atraumatic extraction

Good oral hygiene and periodontal status compatible with socket preservation

Willing and able to attend scheduled follow-up visits and undergo biopsy collection prior to implant placement Able to provide written informed consent

Exclusion Criteria Systemic conditions known to impair bone or soft tissue healing (e.g., uncontrolled diabetes, immunosuppression, osteoporosis)

Current use of medications affecting bone metabolism (e.g., bisphosphonates, corticosteroids, anti-resorptives)

Active periodontal or periapical infection at the extraction site

History of head and neck radiotherapy

Smoking or tobacco use within the past 6 months

Pregnancy or breastfeeding

Known allergy or contraindication to grafting procedures or study-related materials

Inability or unwillingness to comply with follow-up visits or biopsy procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of new bone formation in the extraction socket at 4 months | 4 months after tooth extraction
  Histomorphometric analysis will be performed on biopsies harvested from the preserved sockets. The percentage of newly formed mineralized bone will be calculated as the ratio of new bone area to the total tissue area within the region of interest. Higher values indicate more favorable hard tissue regeneration in the socket preservation site.

SECONDARY OUTCOMES:
Percentage of residual graft material in the extraction socket at 4 months | 4 months after tooth extraction
  Histomorphometric evaluation will quantify the percentage of residual graft material within the preserved socket. The area occupied by residual graft particles will be expressed as a percentage of the total tissue area in the region of interest.
Percentage of new connective tissue in the extraction socket at 4 months | 4 months after tooth extraction
  Histopathological sections will be analyzed to determine the percentage of newly formed connective tissue within the preserved socket. The area of connective tissue will be expressed as a percentage of the total tissue area in the region of interest.
Percentage of newly formed vascularized tissue in the extraction socket at 4 months | 4 months after tooth extraction
  Histomorphometric analysis will assess the proportion of vascularized tissue within the socket. Newly formed vascularized areas will be expressed as a percentage of the total tissue area in the region of interest, reflecting the degree of angiogenesis in the healing socket.
Change in buccolingual ridge width on CBCT from baseline to 4 months | Baseline and 4 months post-extraction
  Standardized cone-beam computed tomography (CBCT) scans will be obtained at baseline (immediately after extraction) and at 4 months. Buccolingual ridge width will be measured at predefined levels, and the change in ridge width over time will be calculated (4 months minus baseline) for each site.
Change in buccal soft tissue thickness measured by intraoral scanner | Baseline and 4 months post-extraction
  Digital intraoral scans will be obtained at baseline and at 4 months. Three-dimensional surface models will be superimposed, and buccal soft tissue thickness at the edentulous ridge will be quantified within a predefined region of interest. The change in thickness will be calculated as the difference between the 4-month and baseline measurements.
Change in width of keratinized mucosa from baseline to 4 months | Baseline and 4 months post-extraction
  The width of keratinized mucosa at the edentulous site will be measured clinically using a periodontal probe at baseline and at 4 months. The change in keratinized mucosa width will be calculated as the difference between the 4-month and baseline measurements.
Change in soft tissue thickness over the preserved socket from baseline to 4 months | Baseline and 4 months post-extraction
  Soft tissue thickness over the preserved socket will be measured using a periodontal probe or standardized transgingival measurement at baseline and at 4 months. The change in soft tissue thickness will be calculated as the difference between the 4-month and baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: okan özen, Principal Investigator — Inonu University Faculty of Dentistry; Arife Sabancı, Study Chair — Inonu University Faculty of Dentistry; Vesile E Toy, Study Chair — Inonu University Faculty of Dentistry
Locations (1):
- Inonu University Faculty of Dentistry, Malatya, Battalgazi-Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The study involves a small, single-center clinical cohort, and the data include identifiable clinical imaging (CBCT scans and intraoral 3-D models) as well as histopathological specimens that cannot be fully anonymized without compromising data integrity. In addition, institutional and national regulations restrict redistribution of such data without additional ethics approval and explicit participant consent.